CLINICAL TRIAL: NCT00638248
Title: International, Multicenter, Double-Blind, Placebo-Controlled, Randomized Phase I/II Trial of Desmoteplase in the Indication of Acute Ischemic Stroke
Brief Title: Dose Escalation of Desmoteplase in Acute Ischemic Stroke (DEDAS)
Acronym: DEDAS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PAION Deutschland GmbH (Industry)
Responsible Party: Karin Wilhelm-Ogunbiyi, MD / Medical Director & Head of Clinical Development, PAION Deutschland GmbH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PN01-CLD-000002/01
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2008-03-19 (Estimated); Status verified 2008-03

CONDITIONS: Stroke
Keywords: Acute ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — salivary plasminogen activator alpha 1, Desmodus rotundus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Desmoteplase 90µg/kg BW
  Interventions: Drug: Desmoteplase
- 2 (Active Comparator): Desmoteplase 125 µg/kg BW
  Interventions: Drug: Desmoteplase
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desmoteplase — Desmoteplase 90µg/kg BW i.v. bolus
  Arms: 1
Drug: Desmoteplase — Desmoteplase 125 µg/kg BW i.v. bolus
  Arms: 2
Drug: Placebo — Placebo i.v. bolus
  Arms: 3

SUMMARY:
The purpose of this study was to explore trends in safety and efficacy, and to find the optimal dose for the subsequent phase III trial. The decision to initiate the phase III trial will depend on both safety (incidence of symptomatic intracranial hemorrhage) and efficacy (reperfusion measured by MRI and correlating with clinical outcome) profiles. The safety (incidence of symptomatic intracranial haemorrhage) and efficacy (reperfusion measured by MRI and correlating with clinical outcome) profiles gained from this study were the basis of planning the phase III.

DETAILED DESCRIPTION:
Acute stroke is the third leading cause of mortality in developed countries and the major medical cause of disability in adults. The outcome can be improved by early treatment with thrombolysis. Alteplase (r-tPA) is the only approved thrombolytic drug in the indication of acute ischemic stroke. However, the use of alteplase is currently restricted by the need to administer it within 3 hours of symptom onset. As the risk of transforming a cerebral infarct into haemorrhage probably rises as the time elapsed increases, a thrombolytic drug that carries a lower risk of haemorrhage than alteplase may offer a wider time-to-treatment window and improve the safety profile.

Desmoteplase (DSPA) with its high fibrin specificity, lack of neurotoxicity, potential neuroprotective effect, non-activation by ß-amyloid, and long terminal half-life may account for an improved safety and efficacy profile within the first 9 hours after onset of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* scoring 4 to 20 on the National Institute of Health Stroke Scale (NIHSS)
* showing a perfusion-diffusion mismatch on MRI of 20 %
* enrolment within a 3 h to 9 h time window after symptom onset.
* 18-85 years of age

Exclusion Criteria:

* Participation in any interventional trial in the previous 30 days.
* Women in the childbearing age.
* Any history of intracranial hemorrhage, subarachnoid hemorrhage, neoplasm, arteriovenous malformation or aneurysm.
* Conditions that, according to the judgment of the investigator, might impose an additional risk to any individual stroke patient when receiving study medication (this applied to patients on platelet-function inhibitors as well).
* MRI exclusion criteria: Evidence of ICH, Evidence of SAH, Signs of extensive early infarction on DWI assessed by evidence of involvement of >1/3 of the middle cerebral artery (MCA) territory. No perfusion deficit, Internal carotid artery (ICA) occlusion ipsilateral to stroke lesion without additional ipsilateral MCA, anterior cerebral artery (ACA) or posterior cerebral artery (PCA) occlusion. Any intracranial pathology that would interfere with the MRI assessment of acute ischemic stroke.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-03; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS), Barthel-Index, mRS | Day 90
Reperfusion after 4-8 h | 8 h
Infarct lesion volume after 30 days | Day 30
Safety & pharmacokinetic outcomes | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Antony J. Furlan, MD, Principal Investigator — Department of Neurology; the Cleveland Clinic Foundation

REFERENCES:
- [Result] Furlan AJ, Eyding D, Albers GW, Al-Rawi Y, Lees KR, Rowley HA, Sachara C, Soehngen M, Warach S, Hacke W; DEDAS Investigators. Dose Escalation of Desmoteplase for Acute Ischemic Stroke (DEDAS): evidence of safety and efficacy 3 to 9 hours after stroke onset. Stroke. 2006 May;37(5):1227-31. doi: 10.1161/01.STR.0000217403.66996.6d. Epub 2006 Mar 30. PMID 16574922
- [Derived] Warach S, Al-Rawi Y, Furlan AJ, Fiebach JB, Wintermark M, Lindsten A, Smyej J, Bharucha DB, Pedraza S, Rowley HA. Refinement of the magnetic resonance diffusion-perfusion mismatch concept for thrombolytic patient selection: insights from the desmoteplase in acute stroke trials. Stroke. 2012 Sep;43(9):2313-8. doi: 10.1161/STROKEAHA.111.642348. Epub 2012 Jun 26. PMID 22738918
- [Derived] Fiebach JB, Al-Rawi Y, Wintermark M, Furlan AJ, Rowley HA, Lindsten A, Smyej J, Eng P, Warach S, Pedraza S. Vascular occlusion enables selecting acute ischemic stroke patients for treatment with desmoteplase. Stroke. 2012 Jun;43(6):1561-6. doi: 10.1161/STROKEAHA.111.642322. Epub 2012 Apr 3. PMID 22474060